CLINICAL TRIAL: NCT03123627
Title: Randomized Clinical Trial, Open, Multicenter Parallel, no Suspension Inferiority Prophylactic Treatment With Valganciclovir in Kidney Transplant CMV-seropositive Cellular Immunity to Develop CD8 + CMV-specific Treatment After Induction Thymoglobulin.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIMOVAL
Record Dates: First submitted 2017-04-19; First posted 2017-04-21 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Kidney Transplant Infection
Keywords: Cytomegalovirus, Seropositive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New profilaxis (Experimental): Prophylaxis is discontinued when the patient developed CMV-specific cellular immunity.
  Interventions: Drug: New profilaxis
- Profilaxis recommended by TTS (Active Comparator): Valganciclovir prophylaxis until day +90 as recommended by the International Consensus document of the TTS.
  Interventions: Drug: Profilaxis recommended

INTERVENTIONS:
Drug: New profilaxis — Primary endpoint: incidence of CMV disease at 12 months after transplantation. Study the predictive value of the assay of CD8 + T cell immunity specific for defined CMV-patients in which they can stop prophylaxis. The definition of CMV disease was based on those recommended by the American Society of Trasnplantation for use in clinical trials (Humar A. Am J Transplant 2006; 6:262-74) criteria.
  Arms: New profilaxis
Drug: Profilaxis recommended — Secondary end points: percentage of patients developing T cell immunity in CMV-specific transplantation after receiving timoglubulina induction and valganciclovir prophylaxis. T cell development inmnunidad CD8 + CMV-specific is defined as production of γ> 0.2 interferon by CD8 + T cells stimulated by CMV-specific CMV antigens (QF reagent).
  Arms: Profilaxis recommended by TTS

SUMMARY:
Hypothesis: Valganciclovir prophylaxis can be discontinued before 3 months in CMV-seropositive renal transplant recipients receiving induction thymoglobulin when developing CMV-specific cellular immunity after transplantation.

Objective Meet the efficacy and safety of valganciclovir prophylaxis suspend in CMV-seropositive kidney transplant recipients with CD8 + cellular immunity CMV-specific transplant, receiving Thymoglobulin induction and maintain cellular immunity-specific CD8 + CMV after transplantation.

Design: noninferiority clinical trial (study A) in CMV-seropositive kidney transplant recipients with CMV-specific cellular immunity pretransplant (Quantiferon reactive CMV) received induction with thymoglobulin

Patients meeting inclusion criteria will be randomized to:

* Control Arm: valganciclovir prophylaxis until day +90 as recommended by the International Consensus document of the TTS (Transplantation 2013:96:333-360).
* Experimental arm: prophylaxis with valganciclovir and determination of CMV-specific cellular immunity day +15, +30, +45 and +60. Prophylaxis was discontinued when the patient developed CMV-specific cellular immunity. Patients who did not develop CMV specific immunity continue prophylaxis until day +90.

Analysis: The incidence of CMV disease according to the strategy used was calculated using Kaplan-Meier curves that were compared using the log-rank test.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant CMV-Seropositive
* CD8+ Tcell CMV especific pretransplant (CMV-reactive quantiferon pretrasplant)
* > 18 years (adult)
* Receiving Thymoglobulin induction therapy
* Receiving Valganciclovir prophylaxis
* Written informed consent for trial entry

Exclusion Criteria:

* Multivisceral transplants including kidney-pancreas.
* HIV-infected Patients
* Patients who can not comply with the monitoring protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence of CMV disease at 12 months after transplantation | 12 months
  Incidence of CMV disease at 12 months after transplantation. Study the predictive value of the assay of CD8 + T cell immunity specific for defined CMV-patients in which they can stop prophylaxis. The definition of CMV disease was based on those recommended by the American Society of Trasnplantation criteria for use in clinical trials

SECONDARY OUTCOMES:
Percentage of patients who recover CMV-specific CD8+ T-cell immunity in the posttransplantation period after receiving thymoglobulin induction therapy and valganciclovir prophylaxis | 12 months
  CMV-specific CD8+ T-cell immunity will be defined using the QF-CMV technique as IFN-γ production equal to or greater than 0.2 IU/mL following stimulation of CD8+ T cells by CMV antigens (QF-CMV "Reactive").CMV replication was considered asymptomatic when it was not accompanied by CMV disease (CMV syndrome or CMV disease)
Incidence of CMV replication | 12 months
  CMV replication was defined as >1500 IU/mL in plasma or >5000 IU/mL in whole blood. CMV replication was considered asymptomatic when it was not accompanied by CMV disease (CMV syndrome or CMV disease)

CONTACTS AND LOCATIONS:
Locations (1):
- Hosìtal Universitario Reina Sofia, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data.
  Who can access the data: Data will be made available only to researchers whose proposed use of the data has been approved by the steering committee.
  Types of analyses: Data will be available for a specified purpose to be communicated in writing to Dr Julián Torre-Cisneros or Dr Sara Cantisán.
  Mechanisms of data availability: Data will be made available only with a signed data access agreement.
  Any additional restrictions: The steering committee has the ultimate decision in approving or denying sample sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning date: 07-01-2021, end date: 30-06-2022
Access Criteria: Data will be made available after the request is approved by the steering committee (J Torre-Cisneros, A Páez-Vega, S Cantisán).
  Requests should be submitted in writing to Dr. Julián Torre-Cisneros (julian.torre.sspa@juntadeandalucia.es) or Dr Sara Cantisán (sacanti@hotmail.com).

REFERENCES:
- [Derived] Paez-Vega A, Gutierrez-Gutierrez B, Aguera ML, Facundo C, Redondo-Pachon D, Suner M, Lopez-Oliva MO, Yuste JR, Montejo M, Galeano-Alvarez C, Ruiz-San Millan JC, Los-Arcos I, Hernandez D, Fernandez-Ruiz M, Munoz P, Valle-Arroyo J, Cano A, Rodriguez-Benot A, Crespo M, Rodelo-Haad C, Lobo-Acosta MA, Garrido-Gracia JC, Vidal E, Guirado L, Cantisan S, Torre-Cisneros J; TIMOVAL Study Group. Immunoguided Discontinuation of Prophylaxis for Cytomegalovirus Disease in Kidney Transplant Recipients Treated With Antithymocyte Globulin: A Randomized Clinical Trial. Clin Infect Dis. 2022 Mar 9;74(5):757-765. doi: 10.1093/cid/ciab574. PMID 34228099